CLINICAL TRIAL: NCT06541652
Title: A French Multicenter Observational Retrospective Study of Rare Primary Liver Cancers
Acronym: FFCD-2205
Status: Recruiting | Type: Observational
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Collaborators: Société Nationale Française de Gastroentérologie (Other)
Responsible Party: Sponsor
Other Study IDs: CAPRIH COHORT; 2023-A01517-38 (Registry Identifier: ID RCB ANSM)
Record Dates: First submitted 2024-07-15; First posted 2024-08-07 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-02

CONDITIONS: Hepatocholangiocarcinoma; Fibrolamellar Carcinoma; Hepatic Epithelioid Hemangioendothelioma; Hepatoblastoma; Hepatic Neuroendocrine Carcinoma; Hepatic Carcinosarcomas; Hepatic Cystadenoma; Hepatic Leiomyosarcomas; Hepatic Angiosarcomas; Cholangiocarcinoma
Keywords: rare primary liver cancers; LIVER; HEPATIC; COHORT; RISK FACTORS
MeSH Terms: conditions — Liver Neoplasms; Fibrolamellar hepatocellular carcinoma; Hepatoblastoma; Cholangiocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — A research blood sample, taken as part of a blood test carried out as part of the patient's care, for living patients with active cancer at the time of registration. If possible, the sample should be taken before a new cancer treatment is carried out.
  The volume of blood collected will be: 2 x 8.5 mL cell free DNA tubes to collect circulating tumor DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of this French multicenter retrospective study is to describ rare primary hepatic cancers clinical, histological and radiological features, to obtain a biological tumor and blood collection, and to evaluate the efficacy of treatments received in clinical practice in order to determine optimal therapeutic sequences. This retrospective cohort will be the backbone of future translational studies aimed at identifying new molecular, histological, circulating and radiological tumor biomarkers, potentially useful at every stage of diagnosis and prognostic or theranostic evaluation.

DETAILED DESCRIPTION:
The aim is to describ rare primary hepatic cancers clinical, histological and radiological features, to obtain a biological tumor and blood collection, and to evaluate the efficacy of treatments received in clinical practice in order to determine optimal therapeutic sequences.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older,
* with histologically proven hepato-cholangiocarcinoma, fibrolamellar hepatocellular carcinoma, epithelioid hemangioendothelioma or hepatic angiosarcoma
* diagnosed after January 01, 2018 living or deceased at the time of registration in the cohort
* for living patients who have not objected to the research: (note of non-objection to be attached° agreeing to participate in ancillary studies must sign the biological consent form for participation in biological studies.

Exclusion Criteria:

* without social security
* No access to tumor block

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the health centers, patients were identified in two ways:
  1. via diagnoses obtained in the anatomopathology departments of each investigating center
  2. via multidisciplinary consultation meetings on primary hepatic tumours/digestive oncology at each investigating center.
  Patients with a diagnosis of rare primary hepatic cancers diagnosed on or after 01/01/2018 may be included, whether alive or deceased at the time of registration in the CAPRIH cohort.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
Description of the clinical, histological and radiological characteristics of various rare primary liver cancers | up to 5 years from the date of diagnosis
  Description of the clinical, histological and radiological characteristics of various rare primary liver cancers

SECONDARY OUTCOMES:
Recurrence-free survival (for non-metastatic patients) | up to 5 years from diagnosis
  Time interval between the date of disease diagnosis and the date of locoregional and/or metastatic recurrence or death (all causes). Patients alive and without recurrence will be censored at the date of last news
Progression-free survival (for metastatic patients) | up to 5 years from diagnosis
  Time interval between the date of diagnosis of the disease and the date of radiological and/or clinical progression or death (all causes). Patients alive and progression-free will be censored at the date of last news.
Overall survival | up to 5 years from diagnosis
  Time interval between the date of diagnosis of the disease and the date of death (from all causes). Living patients will be censored at the date of last news.

CONTACTS AND LOCATIONS:
Overall Officials: jean-charles nault, Pr, Principal Investigator — Federation Francophone de Cancerologie Digestive
Locations (40):
- France (40):
  - CHU Amiens picardie, Amiens
  - Chu Angers, Angers
  - Ch - Centresimone Veil de Beauvais, Beauvais
  - Chu Jean Minjoz, Besançon
  - Ch Bethune Beuvry, Béthune
  - Avicenne, Bobigny
  - Cote de Nacre, Caen
  - Centre Hospitalier, Calais
  - Chu de Clichy Hopital Beaujon, Clichy
  - Centre Hospitalier Universitaire Henri Mondor, Créteil
  - CHU, Dijon
  - Chu Grenobles Alpes, La Tronche
  - Centre Hospital Universitaire de lille, Lille
  - Longjumeau Ch Nord Essone, Longjumeau
  - Ch Edouard Herriot, Lyon
  - Centre Léon Berard, Lyon
  - La Clinique de La Sauvegarde, Lyon
  - Chu Edouard Herriot, Lyon
  - Lyon Cac Leon Berard, Lyon
  - Lyon La Croix Rousse, Lyon
  - Hopital Saint Joseph, Marseille
  - Chu de La Timone, Marseille
  - CHR - Metz Thionville Hopital de Mercy, Metz
  - CHU La Source, Orléans
  - Chu de Paris Saint Antoine, Paris
  - AP - HP - Pitié Salpêtrière, Paris
  - PAU CH, Pau
  - Centre Hospitalier de Perpignan, Perpignan
  - Hopital Haut Leveque, Pessac
  - Chu de Poitiers, Poitiers
  - CH - Annecy Genevois, Pringy
  - Chu Robert Debre, Reims
  - CAC - Eugène Marquis, Rennes
  - Ico Site Rene Gauducheau, Saint-Herblain
  - Hopital Nord Chu Saint Etienne, Saint-Priest-en-Jarez
  - Groupe Hospitalier Rance Emeraude, St-Malo
  - Chu Rangueil, Toulouse
  - Chru de Tours, Tours
  - Chu Paul Brousse, Villejuif
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No